CLINICAL TRIAL: NCT02761668
Title: The Effect of Timing of Orthodontic Therapy on the Outcomes of Regenerative Periodontal Surgery in Patients With Advanced Periodontitis and Pathologic Tooth Migration. A Multi Centre Randomized Clinical Trial.
Brief Title: Timing of Orthodontic Therapy and Regenerative Periodontal Surgery in Advanced Periodontitis Patients With Pathologic Tooth Migration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Karin Jepsen, Associate Professor, University of Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARO/KFO-15-249
Record Dates: First submitted 2016-04-30; First posted 2016-05-04 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Periodontitis; Tooth Migration; Intrabony Periodontal Defect
Keywords: Pathological tooth migration; periodontal regenerative surgery; vertical infrabony defects; xenogeneic bone graft; orthodontic therapy
MeSH Terms: conditions — Periodontitis; Tooth Migration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ParS+Ortho 4W (Experimental): Orthodontic alignment starts 4 weeks post surgical
  Interventions: Procedure: ParS+Ortho 4W
- ParS+Ortho 6M (Active Comparator): Orthodontic alignment starts 6 months post surgical
  Interventions: Procedure: ParS+Ortho 6M

INTERVENTIONS:
Procedure: ParS+Ortho 4W — Orthodontics 4 weeks post surgical
  Arms: ParS+Ortho 4W
Procedure: ParS+Ortho 6M — Orthodontics 6 months post surgical
  Arms: ParS+Ortho 6M

SUMMARY:
Pathologic tooth migration (PTM) is a common complication of advanced periodontitis and often motivation for patients to seek orthodontic therapy. An interdisciplinary approach is required to control the periodontal infection, reconstruct the defects and realign the migrated teeth. The optimal timing of active orthodontics after regenerative therapy is a topic of ongoing debate.

There are no data available from RCTs that have compared the effect of the timing of orthodontic tooth movement (early vs. late) on the outcomes of regenerative periodontal surgery in these patients.

It is the aim of the present randomized clinical multicenter trial to compare 2 different treatment protocols of a combined perio-regenerative and orthodontic therapy in advanced periodontitis patients with intrabony defects and pathologic tooth migration in order to establish whether one treatment modality is superior to the other with regard to clinical outcomes. A total of 46 patients will be enrolled and randomized into 2 treatment groups that differ by the time point of initiation of orthodontic therapy (early: 4 weeks vs. late: 6 months following regenerative periodontal surgery).

Primary outcome measure will be the change in clinical attachment level (CAL gain) at 12 months after regenerative therapy. Secondary outcomes will include changes in probing depth BOP, gingival recession, radiographic bone height and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Advanced periodontitis
* Presence of intrabony defects at a minimum of 2 and a maximum of 7 adjacent teeth (positions 15-25 or 35-45) in either the maxilla or the mandible with PPD of ≥6 mm at a minimum on one site
* Pathologic tooth migration
* Full mouth plaque index (PI) <25% at baseline (after initial non-surgical periodontal therapy)
* Full mouth bleeding on probing (FMBP) <25% at baseline (i.e., following initial non-surgical periodontal therapy)
* Committed to the study and the required follow-up visits

Exclusion Criteria:

Any contraindications for oral surgical procedures

* Uncontrolled diabetes or other uncontrolled systemic diseases
* Disorders or treatments that compromise wound healing
* Medical conditions requiring chronic high dose steroid therapy
* Bone metabolic diseases
* Radiation or other immuno-suppressive therapy
* Infections or vascular impairment at the surgical site
* Presence of oral lesions (such as ulceration, malignancy) or mucosal diseases
* History of malignant disease in the oral cavity or previous radiotherapy to the head
* Inadequate oral hygiene or unmotivated for adequate home care
* Current smokers > 6Cig

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10; Primary Completion 2020-07-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) at test site | 12 months
  Clinical attachment level (CAL)measurements 12 months after surgery

SECONDARY OUTCOMES:
Probing depth (PD) at test site | 24 months
  Probing depth (PD) )measurements 12 and 24 months after surgery
Mean probing depth (PD) | 24 months
  Mean probing depth (PD) )measurements 12 and 24 months after surgery
Bleeding on Probing (BoP) at test site | 24 months
  Bleeding on Probing (BoP) measurements 12 and 24 months after surgery
Mean bleeding on Probing (BoP) | 24 months
  Mean Bleeding on Probing (BoP) measurements 12 and 24 months after surgery
Plaque (PI) at test site | 24 months
  Plaque (PI) measurements 12 and 24 months after surgery
Mean Plaque (PI) | 24 months
  Plaque (PI) measurements 12 months after surgery
Mean clinical attachment level (CAL) | 24 months
  Mean clinical attachment level (CAL)12 months after surgery
PROMS | 24 months
  Patient reported Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Søren Jepsen, Phd, Study Chair — Director; Karin Jepsen, Dr, Principal Investigator — OA; Andreas Jaeger, Phd, Study Chair — Director; Conchita Martin, PhD, Study Chair — Faculty of Odontology, UCM; Mariano Sanz, PhD, Study Chair — Faculty of Odontology, UCM
Locations (2):
- Poliklinik für Parodontologie, Zahnerhaltung und Präventive Zahnheilkunde, Bonn, North Rhine-Westphalia, Germany
- Master de Periodoncia Universidad Complutense, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lindhe J, Svanberg G. Influence of trauma from occlusion on progression of experimental periodontitis in the beagle dog. J Clin Periodontol. 1974;1(1):3-14. doi: 10.1111/j.1600-051x.1974.tb01234.x. No abstract available. PMID 4532114
- [Background] Ericsson I, Thilander B, Lindhe J, Okamoto H. The effect of orthodontic tilting movements on the periodontal tissues of infected and non-infected dentitions in dogs. J Clin Periodontol. 1977 Nov;4(4):278-93. doi: 10.1111/j.1600-051x.1977.tb01900.x. No abstract available. PMID 271655
- [Background] Re S, Corrente G, Abundo R, Cardaropoli D. Orthodontic treatment in periodontally compromised patients: 12-year report. Int J Periodontics Restorative Dent. 2000 Feb;20(1):31-9. PMID 11203546
- [Background] Ghezzi C, Masiero S, Silvestri M, Zanotti G, Rasperini G. Orthodontic treatment of periodontally involved teeth after tissue regeneration. Int J Periodontics Restorative Dent. 2008 Dec;28(6):559-67. PMID 19146051
- [Background] Cardaropoli D, Re S, Manuzzi W, Gaveglio L, Cardaropoli G. Bio-Oss collagen and orthodontic movement for the treatment of infrabony defects in the esthetic zone. Int J Periodontics Restorative Dent. 2006 Dec;26(6):553-9. PMID 17243328
- [Background] Jepsen K, Jaeger A, Jepsen S. Esthetic and functional rehabilitation of a severely compromised central incisor: an interdisciplinary approach. Int J Periodontics Restorative Dent. 2015 May-Jun;35(3):e35-43. doi: 10.11607/prd.2345. PMID 25909531
- [Background] Ghezzi C, Viganò VM, Francinetti P, Zanotti G, Masiero S. Orthodontic treatment after induced periodontal regeneration in deep infrabony defects. Clinical Advances in Periodontics 2013; 3(1), 24-31
- [Background] Cortellini P, Tonetti MS. Clinical concepts for regenerative therapy in intrabony defects. Periodontol 2000. 2015 Jun;68(1):282-307. doi: 10.1111/prd.12048. PMID 25867990
- [Background] Tietmann C, Bröseler F, Axelrad T, Jepsen S. Regenerative procedures and orthodontics in the treatment of severe intrabony defects. A retrospective clinical cohort study. Int Poster J Dent Oral Med 2013; 15 Suppl. Poster 690.
- [Background] Attia MS, Shoreibah EA, Ibrahim SA, Nassar HA. Regenerative therapy of osseous defects combined with orthodontic tooth movement. J Int Acad Periodontol. 2012 Jan;14(1):17-25. PMID 22479985
- [Background] Araujo MG, Carmagnola D, Berglundh T, Thilander B, Lindhe J. Orthodontic movement in bone defects augmented with Bio-Oss. An experimental study in dogs. J Clin Periodontol. 2001 Jan;28(1):73-80. doi: 10.1034/j.1600-051x.2001.280111.x. PMID 11142670
- [Background] Brunsvold MA. Pathologic tooth migration. J Periodontol. 2005 Jun;76(6):859-66. doi: 10.1902/jop.2005.76.6.859. PMID 15948679
- [Background] Cardaropoli D, Gaveglio L, Abou-Arraj RV (2014). Orthodontic movement and periodontal defects: rationale, timing, and clinical implications. Semin Orthod, 20: 177-187.
- [Background] Cortellini P, Stalpers G, Mollo A, Tonetti MS. Periodontal regeneration versus extraction and prosthetic replacement of teeth severely compromised by attachment loss to the apex: 5-year results of an ongoing randomized clinical trial. J Clin Periodontol. 2011 Oct;38(10):915-24. doi: 10.1111/j.1600-051X.2011.01768.x. Epub 2011 Jul 21. PMID 21777268
- [Background] Sanz M, Martin C (2015). Tooth movement in the periodontally compromised patient. In: Clinical periodontology and implant dentistry. Eds: Niklaus P. Lang, Jan Lindhe, pp1297-1324, Wiley
- [Background] Ogihara S, Wang HL. Periodontal regeneration with or without limited orthodontics for the treatment of 2- or 3-wall infrabony defects. J Periodontol. 2010 Dec;81(12):1734-42. doi: 10.1902/jop.2010.100127. Epub 2010 Jul 14. PMID 20629545
- [Background] Re S, Corrente G, Abundo R, Cardaropoli D. Orthodontic movement into bone defects augmented with bovine bone mineral and fibrin sealer: a reentry case report. Int J Periodontics Restorative Dent. 2002 Apr;22(2):138-45. PMID 12019709
- [Derived] Martin C, Tietmann C, Wenzel S, Luengo M, Gaveglio L, Cardaropoli D, Kutschera E, Sanz-Sanchez I, Wullenweber P, Jepsen S, Jepsen K. RCT on orthodontic timing post-periodontal regeneration: root resorption and tooth movement outcomes. Eur J Orthod. 2025 Sep 17;47(5):cjaf078. doi: 10.1093/ejo/cjaf078. PMID 41074768